CLINICAL TRIAL: NCT05137756
Title: Mercuri Analysis Contribution on Handicap Evaluation in ArthrogypOsis, a Congenital Neuromuscular Disease
Acronym: MACHAON
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-MACHAON
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Diagnosis of Arthrogryposis Amyoplasia or Distal Arthrogryposis; 5 Day Multidisciplinary Evaluation in AMC Clinic of the National Reference Center; With Physical Medecin, Medical Genetic and Imaging Departments at the Hospital Grenoble Alpes
Keywords: Arthrogryposis Multiplex Congenita; MRI; mercuri score; fibro-adipous infiltration; fonctionnal capacity; rehabilitation; retrospective observationnal study
MeSH Terms: conditions — Arthrogryposis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Amyoplasia: patient with diagnosis of Amyoplasia
  Interventions: Other: no intervention
- Distal arthrogryposis: patient with diagnosis of Distal arthrogryposis
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The aim is to evaluate the correlation of quantified fibro-adipous infiltration of muscles, using the MRI-based Mercuri score, with deficiencies, activity limitations and social participation in patients with arthrogryposis multiplex congenita.

DETAILED DESCRIPTION:
Arthrogryposis multiplex congenita (AMC) refers to a rare disease spectrum characterized by the presence of joint contractures at birth in at least two different body areas. Causes are multiple. Amyoplasia and distal arthrogryposes are the most frequent causes. Phenotypes consist of muscle weakness and atrophy of variant severity and joint deformities. The impact on mobility, activities or daily living and participation is variable (Dai et al, 2018).

Mercuri et al. (Mercuri et al, 2002) have developed a semi-quantitative score to mesure fibro-adipous muscle infiltration on muscle MRI.

Correlations between fibro-adipous infiltration and muscular deficits have already been studied in other neuromusclar diseases such as Pompe disease (Figueroa-Bonaparte et al, 2016) or Duchenne muscular dystrophy (Brogan et al, 2018). These studies revealed good correlation between disease onset, muscle strength and the degree of muscle fibro-adipous infiltration, calculated using the Mercuri score. The authors concluded that muscular MRI can be used to follow the neuromuscular disease progression as it is correlated with muscle function.

Contrary to these progressive diseases, AMC is a congenital non progressive condition. It is therefore tempting to hypothesize that the muscular fibro-adipous infiltration in these patients could be of prognostic value for future capacities.

Our aim is to evaluate the fibro-adipous muscle infiltration in a thoroughly phenotyped cohort of adult patients with Amyoplasia and Distal Arthrogryposes using the Mercuri score, based on muscular MRI, in order to evaluate the correlation with deficiencies, activity limitations and social participation.

ELIGIBILITY:
Inclusion Criteria:

* adults
* with a diagnostic of Amyoplasia or distal arthrogryposis
* evaluated by a all body MRI
* functionnal evaluation during day hospitalisation in neurorehabilitation department
* between 2010 and october 2020

Exclusion Criteria:

* other aetiology of Arthrogryposis multiplex congenita (AMC)
* incomplete MRI or medical files
* interaction with other disease

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adults with a diagnostic of Amyoplasia or distal arthrogryposis, evaluated by a all body MRI, and functionnal evaluation during day hospitalisation in adult neurorehabilitation department of grenoble, between 2010 and october 2020
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Mercuri Scores of upper limbs, lower limbs,and trunk evaluated on MRI T1 | during 5 day evaluation
  The degree of muscle fat infiltration was assessed with at least 2 visible slices. We used the four-point scale proposed by Mercuri et al 2002. Each muscle was staged as follows: 1. Normal appearance, 2. Mild involvement. 3. Moderate involvement. 4. Severe involvement.

SECONDARY OUTCOMES:
muscle weakness | during 5 day evaluation
  muscular weakness was assessed by function (flexion, extension etc.) and not by each muscle, using the Medical Research Council scale (0-5) for muscle weakness. The grading was as follows: 0, no contraction; 1, flicker or trace of contraction; 2, active movement possible only with gravity eliminated; 3, active movement against gravity in the whole range of motion; 4, active movement against gravity and resistance; 5, quasi-normal strength.
passive range of motion | during 5 day evaluation
  passive range of motion evaluated by physiotherapists, The range of motion of each movement (i.e. amplitude) was normalized with respect to the normal maximal movement, expressed as percentages
6 minutes walking test | during 5 day evaluation
  Mobility was assessed by the 6MWT20, performed by individuals who were asked to walk as self-preferred speed in a straight line on the floor with sequences of 30 meters, with a half-turn at each end. In case of interruption (fatigue, pain, dyspnea), patients were allowed to rest, until they felt able to restart.
reaching score | during 5 day evaluation
  The ability to reach some body targets with upper limbs was assessed by ad hoc test. Individuals sitting on a chair were instructed to successively touch their mouths, heads, necks, backs, opposite shoulders, ipsilateral shoulders, knees and feet, with both hands. Each successful touch scored two points if easily performed, and one point if performed with difficulty. The total score was calculated on both sides averaged and ranged from 0 to 16 points.
Functionnal independance measure | during 5 day evaluation
  Designed to assess areas of dysfunction in activities that commonly occur in subjects with any progressive, reversible or stable neurologic, musculoskeletal, or other disorder ie patients with functional mobility impairmentsThe motor subscale includes: Eating, Grooming, Bathing, Dressing, upper body, Dressing, lower body, Toileting, Bladder management, Bowel management, Transfers - bed/chair, wheelchair, Transfers - toilet, Transfers - bath/shower, Walk/wheelchair, Stairs, The cognition subscale includes: Comprehension, Expression, Social interaction, Problem solving, Memory Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item
pain evaluation | during 5 day evaluation
  based on patient declaration, absence or presence (with pain scale) and pain localisations
activities in daily life | during 5 day evaluation
humain and technical aid | during 5 day evaluation
  utilisation of technical aid (walking stick, manual or electric wheelchair), or humain for daly life activities
respiratory and speech difficulties | during 5 day evaluation
  surgical history, capacity to speech
surgical history | during 5 day evaluation
  personnal surgical history for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Dominic PERENNOU, MDPHD, Study Director — CHU Grenoble Alpes; Klaus DIETERICH, MD, Study Director — CHU Grenoble Alpes
Locations (1):
- Chu Grenoble Alpes, La Tronche, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu CY, Yao J, Kovacs WC, Shrader JA, Joe G, Ouwerkerk R, Mankodi AK, Gahl WA, Summers RM, Carrillo N. Skeletal Muscle Magnetic Resonance Biomarkers in GNE Myopathy. Neurology. 2021 Feb 2;96(5):e798-e808. doi: 10.1212/WNL.0000000000011231. Epub 2020 Nov 20. PMID 33219145
- [Result] Hall JG. Arthrogryposis multiplex congenita: etiology, genetics, classification, diagnostic approach, and general aspects. J Pediatr Orthop B. 1997 Jul;6(3):159-66. PMID 9260643
- [Result] Mercuri E, Pichiecchio A, Counsell S, Allsop J, Cini C, Jungbluth H, Uggetti C, Bydder G. A short protocol for muscle MRI in children with muscular dystrophies. Eur J Paediatr Neurol. 2002;6(6):305-7. doi: 10.1016/s1090-3798(02)90617-3. PMID 12401454
- [Result] Figueroa-Bonaparte S, Segovia S, Llauger J, Belmonte I, Pedrosa I, Alejaldre A, Mayos M, Suarez-Cuartin G, Gallardo E, Illa I, Diaz-Manera J; Spanish Pompe Study Group. Muscle MRI Findings in Childhood/Adult Onset Pompe Disease Correlate with Muscle Function. PLoS One. 2016 Oct 6;11(10):e0163493. doi: 10.1371/journal.pone.0163493. eCollection 2016. PMID 27711114
- [Result] Dai S, Dieterich K, Jaeger M, Wuyam B, Jouk PS, Perennou D. Disability in adults with arthrogryposis is severe, partly invisible, and varies by genotype. Neurology. 2018 May 1;90(18):e1596-e1604. doi: 10.1212/WNL.0000000000005418. Epub 2018 Apr 6. PMID 29626181